CLINICAL TRIAL: NCT00000774
Title: A Phase I Study to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Antigen in Children Born to HIV-Infected Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry); Biocine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 230; 11207 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; Virus Replication; HIV Envelope Protein gp120; AIDS Vaccines; HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Patients who will receive rgp120/HIV-1MN
  Interventions: Biological: rgp120/HIV-1MN
- 2 (Experimental): Patients who will receive rgp120/HIV-1SF2
  Interventions: Biological: rgp120/HIV-1 SF-2
- 3 (Placebo Comparator): Patients who will receive the placebo counterpart of 120/HIV-1MN
  Interventions: Biological: Placebo version of rgp120/HIV-1MN
- 4 (Placebo Comparator): Patients who will receive the placebo counterpart of rgp120/HIV-1SF2
  Interventions: Biological: Placebo version of rgp120/HIV-1SF2

INTERVENTIONS:
Biological: rgp120/HIV-1MN — Administered at weeks 0, 4, 8, 12, and 20. Individual group assignment will determine specific dosage and schedule.
  Arms: 1
Biological: rgp120/HIV-1 SF-2 — Administered at weeks 0, 4, 8, 12, and 20. Individual group assignment will determine specific dosage and schedule.
  Arms: 2
Biological: Placebo version of rgp120/HIV-1MN — Administered at weeks 0, 4, 8, 12, and 20. Individual group assignment will determine specific dosage and schedule.
  Arms: 3
Biological: Placebo version of rgp120/HIV-1SF2 — Administered at weeks 0, 4, 8, 12, and 20. Individual group assignment will determine specific dosage and schedule.
  Arms: 4

SUMMARY:
PRIMARY: To determine the safety of envelope recombinant proteins rgp120/HIV-1MN (Genentech) and rgp120/HIV-1SF2 (Chiron/Biocine) in infants who are of indeterminate HIV status born to HIV-infected women. To evaluate changes in viral load in infants proven to be infected and absolute CD4 counts in all immunized infants.

SECONDARY: To evaluate the immunogenicity of these envelope recombinant proteins in infants of indeterminate HIV status born to HIV-infected women.

Only 30-50 percent of HIV-infected infants have detectable virus at birth. Successful early sensitization to HIV envelope epitopes may help prevent infection or, alternatively, may enhance HIV-specific immune function to alter HIV replication and disease progression.

DETAILED DESCRIPTION:
Only 30-50 percent of HIV-infected infants have detectable virus at birth. Successful early sensitization to HIV envelope epitopes may help prevent infection or, alternatively, may enhance HIV-specific immune function to alter HIV replication and disease progression.

Newborns are randomized to one of three different doses of either rgp120/HIV-1MN or rgp120/HIV-1SF2 or their matching placebos. At each dose level, 12 patients receive vaccine and three patients receive placebo. Immunizations are performed at 0, 4, 12, and 20 weeks, and patients are followed until 2 years of age. Three of four patients treated at a given dose level must have received two immunizations without evidence of grade 3 or 4 clinical or laboratory toxicity before dose escalation occurs. Twelve additional patients are treated with the optimal dose of each vaccine at weeks 0, 2, 8, and 20 (An accelerated schedule PER AMENDMENT 3/20/96. Changed from - 0, 4, 8, and 20) accompanied by three additional placebo patients per vaccine. PER AMENDMENT 3/20/96: The optimal dose of rgp120/HIV-1MN is 100 mcg and will be given to the 12 patients and the placebo will be given to 3. The optimal dose of rgp120/HIV-1SF2 is 5 mcg and will be given to the 12 patients and the placebo will be given to 3.

PER 2/3/95 AMENDMENT: After the initial patients are enrolled, 18 additional newborns will be randomized to one of the three dose levels of rgp120/HIV-1MN (with no placebos). PER AMENDMENT 6/5/95: Another group of 18 newborns will be randomized to one of three treatments representing 3 different doses of the Chiron/Biocine vaccine (with no placebos).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Coenrollment in a therapeutic protocol if begun at least 30 days following the week 20 immunization.
* Routine immunizations if given more than 1 week before or after study vaccine.

Patients must be:

* > 37 weeks gestation and < 72 hours of age born to HIV-infected women.
* NOT born to women who received either passive or active immunotherapy during pregnancy.
* NOT breast-fed.
* NOT born to women who are hepatitis B surface antigen positive.
* Receiving AZT at study entry (except infants enrolled in ACTG 076).

NOTE:

* Parent or guardian must provide informed consent and be willing to comply with study requirements.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Documented or suspected serious bacterial infection, metabolic illness, or other immediate life-threatening conditions.

Concurrent Medication:

Excluded:

* Passive or active HIV-specific immunotherapy other than the study candidate vaccines.
* Investigational medications.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Study Completion 1999-01 (Actual)

PRIMARY OUTCOMES:
Development of adverse clinical, laboratory, or immunological responses to any of the recombinant vaccines | Throughout study
Changes in viral load in infants found to be HIV infected | Throughout study
Changes in the slope of absolute CD4 counts in all immunized children | Throughout study

SECONDARY OUTCOMES:
Changes in immune response to the vaccine candidates | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Borkowsky W, Study Chair — NYU MEDICAL CENTER; Wara DW, Study Chair — UCSF Moffit Hospital
Locations (37):
- United States (36):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - San Francisco Gen. Hosp., San Francisco, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane Univ. Health Science Ctr., Tulane Univ. Hosp. & Clinic, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Brigham and Women's Hosp., Div. of Infectious Disease, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - NJ Med. School CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Hosp. of the Univ. of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
  - UW School of Medicine - CHRMC, Seattle, Washington
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Rogers MF, Mofenson LM, Moseley RR. Reducing the risk of perinatal HIV transmission through zidovudine therapy: treatment recommendations and implications. J Am Med Womens Assoc (1972). 1995 May-Aug;50(3-4):78-82, 93. PMID 7657952
- [Background] Cunningham CK, Wara DW, Kang M, Fenton T, Hawkins E, McNamara J, Mofenson L, Duliege AM, Francis D, McFarland EJ, Borkowsky W; Pediatric AIDS Clinical Trials Group 230 Collaborators. Safety of 2 recombinant human immunodeficiency virus type 1 (HIV-1) envelope vaccines in neonates born to HIV-1-infected women. Clin Infect Dis. 2001 Mar 1;32(5):801-7. doi: 10.1086/319215. Epub 2001 Feb 28. PMID 11229849
- [Background] Borkowsky W, Wara D, Fenton T, McNamara J, Kang M, Mofenson L, McFarland E, Cunningham C, Duliege AM, Francis D, Bryson Y, Burchett S, Spector SA, Frenkel LM, Starr S, Van Dyke R, Jimenez E. Lymphoproliferative responses to recombinant HIV-1 envelope antigens in neonates and infants receiving gp120 vaccines. AIDS Clinical Trial Group 230 Collaborators. J Infect Dis. 2000 Mar;181(3):890-6. doi: 10.1086/315298. PMID 10720509